CLINICAL TRIAL: NCT06041165
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Kinetic Effects in Healthy Volunteers With Normal or Mildly Elevated Triglycerides
Brief Title: A Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of JS401
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: JS401-001
Record Dates: First submitted 2023-09-01; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: JS401 injection (Experimental)
  Interventions: Drug: JS401
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JS401 — Single dose of JS401 by subcutaneous (sc) injections
  Arms: Experimental: JS401 injection
Drug: Placebo — Calculated volume to match active treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetcs and pharmacodynamics of single-dose of JS401 in healthy volunteers with normal or mildly elevated triglycerides.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18~60 (inclusive) at the time of signing the ICF, with no less than 1/3 of either gender;
2. Fasting TG≥1.1mmol/L (100 mg/dL) and ≤ 5.0mmol/L (450mg/dL) at screening; (3) Fasting LDL-C at screening> 1.8 mmol/L (70 mg/dL).

Exclusion Criteria:

1. Have a medical history or clinical evidence that the subject has obvious concomitant diseases (including but not limited to: cardiovascular, respiratory, digestive, urinary, neurological, blood, immunological, endocrine and metabolic, infection, etc.), or any clinically significant abnormalities found in physical examination, laboratory examination, and ECG examination, which are judged by the investigator to not meet the standards of clinical health or are not suitable for participating in clinical trials;
2. Acute or chronic infection requiring hospitalization or undergoing systemic parenteral therapy (antiviral/bacterial/fungal/parasitic, etc.) within 60 days prior to randomization;
3. Positive for syphilis antibodies, or positive for human immunodeficiency virus (HIV) antibodies, or positive for hepatitis C virus (HCV) antibodies, or positive for hepatitis B virus surface antigen (HBsAg) at screening;
4. History of substance abuse within 12 months prior to screening, or positive urine drug screening at screening;
5. History of alcohol dependence within 6 months prior to screening, or positive breath test for alcohol at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-06-29 (Estimated); Study Completion 2024-09-21 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 112 days post-dose
  Number of Participants with Adverse Events (AEs)

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Up to 48 hours post-dose
  Peak Plasma Concentration of JS401
Time to Maximum Plasma Concentration (Tmax) | Up to 48 hours post-dose
  Time to Maximum Plasma Concentration of JS401
Terminal Elimination Half-Life (t1/2) | Up to 48 hours post-dose
  Terminal Elimination Half-Life (t1/2) of JS401
Area Under the Plasma Concentration Versus Time Curve (AUC) | Up to 48 hours post-dose
  Area Under the Plasma Concentration Versus Time Curve of JS401
Angiopoietin-like 3 (ANGPTL3) | Up to 112 days post-dose
  Reduction in Fasting Serum ANGPTL3 from Pre-Dose Baseline
Triglycerides | Up to 112 days post-dose
  Reduction in Fasting Serum LDL-C from Pre-Dose Baseline
immunogenic characteristics ADA of JS401 | Up to 112 days post-dose
  The number and percentage of subjects who were positive for anti-JS401 anti-drug antibody (ADA) after administration of JS401 injection were counted, and the titer of ADA-positive samples was analyzed.
Low-density lipoprotein cholesterol (LDL-C) | Up to 112 days post-dose
  Reduction in Fasting Serum LDL-C from Pre-Dose Baseline
Non-high-density lipoprotein cholesterol (non-HDL-C) | Up to 112 days post-dose
  Reduction in Fasting Serum non-HDL-C from Pre-Dose Baseline
Very low-density lipoprotein cholesterol (VLDL-C) | Up to 112 days post-dose
  Reduction in Fasting Serum VLDL-C from Pre-Dose Baseline
High-density lipoprotein cholesterol (HDL-C) | Up to 112 days post-dose
  Reduction in Fasting SerumHDL-C from Pre-Dose Baseline
Lipoprotein (a) (Lp(a)) | Up to 112 days post-dose
  Reduction in Fasting Lp(a) from Pre-Dose Baseline
Apolipoprotein B (ApoB) | Up to 112 days post-dose
  Reduction in Fasting ApoB from Pre-Dose Baseline
Apolipoprotein A1 (ApoA1) | Up to 112 days post-dose
  Reduction in Fasting ApoA1 from Pre-Dose Baseline
Q-T interval | Up to 112 days post-dose
  Change in QTc from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No